CLINICAL TRIAL: NCT01538355
Title: A Randomised Controlled Pilot Study to Compare the Effects of Prolonged Fasting and Ketogenic Low Glycemic Load Treatment on Health Related Quality of Life in Relapsing-remitting Multiple Sclerosis.
Brief Title: A Pilot Trial to Test the Feasibility of Prolonged Fasting and Ketogenic Diet in Relapsing-remitting Multiple Sclerosis
Acronym: IGEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Markus Bock, MD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGEL
Record Dates: First submitted 2012-02-15; First posted 2012-02-24 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: multiple sclerosis; diet; prolonged fasting; caloric restriction; ketogenic low glycemic load treatment; health related quality of life; ketogenic diet; neurodegeneration; neuroinflammation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Nerve Degeneration; Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prolonged fasting (Experimental): Patients undergo an initial 7-day fasting episode.
  Interventions: Other: Prolonged Fasting
- Ketogenic low glycemic load treatment (Experimental): Patients receive a ketogenic low glycemic load treatment from the outset of the study.
  Interventions: Other: Ketogenic low glycemic load treatment
- Control diet (Experimental): Patients stay on their regular diet.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Prolonged Fasting — Patients enhance their regular diet with an initial 7-day fasting episode.
  Arms: Prolonged fasting
Other: Ketogenic low glycemic load treatment — 6 months of ketogenic low glycemic load treatment from the study outset.
  Arms: Ketogenic low glycemic load treatment
Other: Control diet — Patients stay on their regular diet.
  Arms: Control diet

SUMMARY:
It is well accepted that nutrition as an environmental factor is involved in the pathogenesis of multiple sclerosis. But is there a role for prolonged fasting and ketogenic low glycemic load treatment to alter the course of multiple sclerosis (MS)? The investigators think yes there is. Primarily the investigators want to detect if these diets are feasible for MS patients. Therefore the investigators examine the impact of this dietary intervention on the health related quality of life for individuals after 7 days, 3 months and 6 months in compare to baseline. Secondarily the investigators focus on endocrinological and immunological changes after 7 days, 3 months and 6 months in compare to baseline.

DETAILED DESCRIPTION:
In this controlled randomised pilot study the patients are allocated to 1. a ketogenic low glycemic load treatment from the outset of the study for 24 weeks or 2. enhance their regular diet with an initial 7-day fasting followed by a Mediterranean diet pattern until the study end or 3. stay on their regular diet (control group) from the outset of the study for 24 weeks. The investigators will then assess the differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS
* Stable immunomodulatory treatment or no treatment at least 6 months prior to inclusion
* Expanded disability status scale < 7
* Body mass index (BMI) > or = 18,5 OR BMI > or = 45 with no risk factors
* Not pregnant or breast-feeding
* No serious mental health illness such as dementia or schizophrenia;
* No use of a weight loss therapy in the month prior to screening.

Exclusion Criteria:

* Start or changes if immunomodulatory treatment < 7 months prior to screening
* SPMS or PPMS
* Relapse or corticosteroid use < 30 days prior to screening
* Diabetes or any metabolic defects
* Bulimia
* Anorexia
* Drug abuse

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-07-30 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Multiple Sclerosis Quality of Life-54 questionnaire: Proof of feasibility at 6 months. | Visit: Baseline, month 1, month 3 and month 6
  Two summary scores: physical health und mental health, 12 subscales and 2 single item scales.

SECONDARY OUTCOMES:
Adherence rates, number of participants with adverse events and laboratory parameters at 6 months. | Visits: Baseline, month 1, month 3 and month 6
  Multiple sclerosis functional composite; fatigue scores, body composition; body weight; lipid profile, liver enzymes, insulin, glucagon

CONTACTS AND LOCATIONS:
Overall Officials: Markus Bock, MD, Principal Investigator — Charité-Universitätsmedizin Berlin, Berlin Germany
Locations (1):
- Charité-Universitätsmedizin, Berlin, Germany

REFERENCES:
- [Background] Piccio L, Stark JL, Cross AH. Chronic calorie restriction attenuates experimental autoimmune encephalomyelitis. J Leukoc Biol. 2008 Oct;84(4):940-8. doi: 10.1189/jlb.0208133. Epub 2008 Aug 4. PMID 18678605
- [Background] Kim DY, Hao J, Liu R, Turner G, Shi FD, Rho JM. Inflammation-mediated memory dysfunction and effects of a ketogenic diet in a murine model of multiple sclerosis. PLoS One. 2012;7(5):e35476. doi: 10.1371/journal.pone.0035476. Epub 2012 May 2. PMID 22567104
- [Result] Swidsinski A, Dorffel Y, Loening-Baucke V, Gille C, Goktas O, Reisshauer A, Neuhaus J, Weylandt KH, Guschin A, Bock M. Reduced Mass and Diversity of the Colonic Microbiome in Patients with Multiple Sclerosis and Their Improvement with Ketogenic Diet. Front Microbiol. 2017 Jun 28;8:1141. doi: 10.3389/fmicb.2017.01141. eCollection 2017. PMID 28702003
- [Derived] Bock M, Steffen F, Zipp F, Bittner S. Impact of Dietary Intervention on Serum Neurofilament Light Chain in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2021 Nov 11;9(1):e1102. doi: 10.1212/NXI.0000000000001102. Print 2022 Jan. PMID 34764215
- [Derived] Bock M, Karber M, Kuhn H. Ketogenic diets attenuate cyclooxygenase and lipoxygenase gene expression in multiple sclerosis. EBioMedicine. 2018 Oct;36:293-303. doi: 10.1016/j.ebiom.2018.08.057. Epub 2018 Oct 3. PMID 30292675
- [Derived] Choi IY, Piccio L, Childress P, Bollman B, Ghosh A, Brandhorst S, Suarez J, Michalsen A, Cross AH, Morgan TE, Wei M, Paul F, Bock M, Longo VD. A Diet Mimicking Fasting Promotes Regeneration and Reduces Autoimmunity and Multiple Sclerosis Symptoms. Cell Rep. 2016 Jun 7;15(10):2136-2146. doi: 10.1016/j.celrep.2016.05.009. Epub 2016 May 26. PMID 27239035